CLINICAL TRIAL: NCT06069167
Title: Bowel Urgency in Inflammatory Bowel Disease
Acronym: URGENT-1
Status: Completed | Type: Observational
Sponsor: Paris IBD Center (Other)
Responsible Party: Sponsor
Other Study IDs: PIBDC-2023-01
Record Dates: First submitted 2023-10-01; First posted 2023-10-05 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
Keywords: Bowel urgency; URGENT index; IBD; UNRS (Urgency Numeric Rating Scale); GVE (Global Visual Evaluation)
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Collection of data related to bowel urgency — Data will be extracted from the patient's medical record and patients will be interviewed to collect data specific to the research

SUMMARY:
Bowel urgency is commonly defined as the sudden need to rush to the bathroom to empty one's bowel. In the field of inflammatory bowel disease (IBD) (including Crohn's disease (CD) and ulcerative colitis (UC)), bowel urgency is part of the top five research priorities for future IBD nursing research, and it is a symptom that patients consider to be most important when prioritizing their disease control. Urgency is a patient-reported outcome associated with compromised quality of life and future risk of hospitalizations, corticosteroids, and colectomy in patients with UC.

A meta-analysis of 321 studies examining bowel urgency revealed that only one-third of these clinical studies clearly defined the concept of bowel urgency. Definition of bowel urgency was heterogeneous as 14 different definitions were identified. In most of these studies, non-validated questionnaires were used. They are based on subjective responses of the patients, and they could determine evaluation bias. These data emphasize the lack of standardization in bowel urgency assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged at least 18 years old
* Diagnosis of inflammatory bowel disease according to the European Crohn´s and Colitis Organisation criteria for at least 3 months
* Person who has received full information about the organization of the research and who has not objected to his or her participation and to the use of his or her data
* Person affiliated to or beneficiary of a social security plan

Exclusion Criteria:

* Person unable to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inflammatory bowel disease patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Prevalence of bowel urgency in a cohort of patients with inflammatory bowel disease | Through study completion, an average of 12 months
  Inability to defer defecation for more than 15 minutes in patients with inflammatory bowel disease

SECONDARY OUTCOMES:
Prevalence of bowel urgency in a cohort of Crohn's disease patients | Through study completion, an average of 12 months
  Inability to defer defecation for more than 15 minutes in patients with Crohn's disease
Prevalence of bowel urgency in a cohort of ulcerative colitis patients | Through study completion, an average of 12 months
  Inability to defer defecation for more than 15 minutes in patients with ulcerative colitis
Development of the URGENT index (i.e. inflammatory bowel disease-specific bowel urgency index) | Through study completion, an average of 12 months
  Components of the index based on variables describing in systematic review Caron B et al. Clin Gastroenterol Hepatol. 2023 and IBD expert opinion
To identify IBD-related risk factors associated with an increased risk of bowel urgency | Through study completion, an average of 12 months
  Inability to defer defecation for more than 15 minutes and potentially predictive factors (i.e. baseline characteristics)
Correlation between the URGENT index and the Urgency Numeric Rating Scale | Through study completion, an average of 12 months
  Relationships between changes in the URGENT index and changes in the Urgency Numeric Rating Scale
Correlation between the URGENT index and a Global Visual Evaluation | Through study completion, an average of 12 months
  Relationship between changes in the URGENT index and changes in the Global Visual Evaluation on a 10-point visual analog scale ranging from 0 (minimal activity) to 10 (maximal activity)
Most appropriate definition of bowel urgency for patients with IBD | Through study completion, an average of 12 months
  Urgent desire to defecate and/or extreme desire to defecate and/or immediate need to defecate and/or inability to defer defecation for more than 2 minutes and/or inability to defer defecation for more than 5 minutes and/or inability to defer defecation for more than 20 minutes and/or inability to defer defecation for more than 30 minutes and/or having to rush to the toilet and/or not making it to a toilet in time and/or having to stop whatever to have a bowel movement and/or difficult to withstand urge to open bowels and/or running to the bathroom and/or inability to delay bowel movements

CONTACTS AND LOCATIONS:
Locations (1):
- Institut des MICI, Neuilly-sur-Seine, France